CLINICAL TRIAL: NCT01182506
Title: Rehabilitation of Cognitive Changes in Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MARTELL FOUNDATION (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-105
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Cogmed Working Memory Training (CWMT); cognitive; 10-105; Breast cancer survivor
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- Breast cancer survivors (Experimental): Participants from both groups will be asked to complete two follow up neurocognitive assessments face to face at MSKCC. The first will be completed within 1-4 weeks after completing the memory training and the second will take place 3-4 months after completing the memory training. Collateral sources will be contacted at these same points to complete their brief assessments as well to test for maintenance of the treatment effect.
  Interventions: Behavioral: Cogmed Working Memory Training Program
- Collateral source (Experimental): Participants from both groups will be asked to complete two follow up neurocognitive assessments face to face at MSKCC. The first will be completed within 1-4 weeks after completing the memory training and the second will take place 3-4 months after completing the memory training. Collateral sources will be contacted at these same points to complete their brief assessments as well to test for maintenance of the treatment effect.
  Interventions: Behavioral: Cogmed Working Memory Training Program

INTERVENTIONS:
Behavioral: Cogmed Working Memory Training Program — Women will be randomized to one of two 5-week rehabilitation software training programs that train working memory called Cogmed Working Memory Training Program.
  The training software will be provided to each participant. For each group, training occurs for 30 minutes a day, 5 days a week for 5 weeks. As part of the set-up, training data is uploaded to the internet at a minimum of every 3 days. This function allows the "coach" (in this case, the PI and RSA) to review the training. A weekly "coach" phone call is made to review the training results, answer questions, troubleshoot, and motivate the participant. Participants can load the software onto multiple computers to provide flexibility for them to do training at home, after work, when they are away from home.

SUMMARY:
The purpose of this study is to test a memory training program for breast cancer survivors who have problems with memory after receiving chemotherapy. Since breast cancer survivors have been reported to have trouble with their memory, a program to help these problems is important. Studies have shown that a 5-week software training program improved memory in pediatric cancer survivors and other disorders like stroke, but it has not been tested for breast cancer survivors. This study will see if breast cancer survivors can improve their memory and attention problems by using either one of two software versions of the program. One version is called Cogmed Working Memory Training, and the other is a comparison version of the software that has the same exercises but is less difficult. People who decide to participate in the study will be randomly given one of the two versions.

ELIGIBILITY:
Note: Any participant who reports tics can be included, however participants will be told tics may increase during the training period.

Inclusion Criteria:

Patients

* Female breast cancer survivors who have received adjuvant chemotherapy 1-10 years from the time of recruitment either at MSKCC or elsewhere
* Stage I, II, III breast cancer as noted in pathology reports or by clinician judgement.
* No evidence of disease at time of screening
* Age range 18 years old through <70 years old
* Must be able speak, read and write English well enough to complete written and verbal assessments and neurocognitive tests. The software was developed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures.
* Must demonstrate cognitive deficiency, which is defined as 1.0 standard deviations below normative data on at least one of the pre-screen phone assessments (WAIS-III Digit Span, Symbol Digit Modalities Test, Controlled Oral Word Association Test, Rey Auditory Verbal Learning Test) or must have 1.0 standard deviations difference from the pre-morbid estimate of cognitive functioning, Wide Range Achievement Test 4: Reading subtest, and one of the pre-screen phone assessment measures.
* Must have basic computer skills such as able to turn on a computer, open the program, login, and use a mouse.
* Participants must have the ability to upload their data via the internet. A study laptop can be loaned out to participants who do not have a computer or the appropriate operating systems.

Collateral Participant (if such person is available to the participant, not a requirement of the study) Family member or friend (i.e., collateral) identified by a patient who has at least weekly face to face contact with the patient

* Collateral person is at least 18 years of age
* Family member or friend has adequate English fluency for completion of data collection. The surveys were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures.
* Able to provide informed consent

Exclusion Criteria:

Patients

* History of neurological disorder with cognitive symptoms (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis, seizure disorder) as per self report or as documented in the electronic medical record.
* History of mental retardation, learning disorder bipolar disorder, schizophrenia, substance use disorder(s), or uncontrolled depression as per self report or as documented in the medical record.
* History of Traumatic Brain Injury with > or = to 30 minutes loss of consciousness or cognitive sequelae as per self report or as documented in the medical record.
* History of Stroke as per self report or as documented in the medical record.
* Prior history or secondary diagnosis of other cancers except for basal cell carcinoma or melanoma treated with surgery only
* History of multiple courses of chemotherapy.
* Evidence of recurrence at time of screening
* A hearing or visual deficit that impairs the ability to use the software.
* Significant cognitive or psychiatric disturbance sufficient, in the investigator's judgment, to preclude providing informed consent.
* Males will be excluded as only a minority of men gets breast cancer. Thus, there would not be enough men to have equivalent groups to statistically control for possible gender effects.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of working memory training | 2 years
  in breast cancer survivors based on improved performance on neuropsychological tests of working memory.

SECONDARY OUTCOMES:
Test whether or not working memory training in breast cancer survivors is associated with greater gains in the software's "Improvement Index". | 2 years
Investigate whether breast cancer survivors perceive functional improvement following working memory training. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ryan, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm